CLINICAL TRIAL: NCT00270725
Title: The Effectiveness of Antiretroviral Therapy in Reducing the Costs of HIV/AIDS
Brief Title: Impact of Anti-HIV Treatment on Labor Productivity and Costs in South Africa
Status: Withdrawn | Type: Observational
Why Stopped: Enrollment never initiated, study withdrawn.
Sponsor: Boston University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sydney Rosen, Boston University
Other Study IDs: RTC-BU-01
Record Dates: First submitted 2005-12-27; First posted 2005-12-28 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; Labor productivity; Antiretroviral therapy; South Africa
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to determine the impact of anti-HIV treatment on the work attendance of employed people in South Africa. The study will enroll participants from a large manufacturing and distribution firm in South Africa.

DETAILED DESCRIPTION:
Little is known about the economic benefits of providing antiretroviral therapy (ART) for HIV infected patients in sub-Saharan Africa and other resource-limited areas. In South Africa, an increasing number of private sector firms are providing access to ART for their employees. One of the barriers to such action, however, is the lack of available information on the success of ART in restoring workers to full productivity, retaining skilled employees in the workforce, and reducing the costs of medical care and death and disability benefits. HIV infected employees on ART may be absent from work less often than untreated HIV infected employees, but more often than HIV uninfected employees. This study will collect data from an independent HIV/AIDS disease treatment program and a large private sector employer in Johannesburg, South Africa to estimate the benefits and costs for businesses to provide ART to eligible employees.

The study will combine individual-level medical outcome and treatment cost data from the treatment program with data on employee work attendance and retention in the workforce from the participating employer. The work attendance of HIV infected employees enrolled in the HIV/AIDS treatment program (index participants) who are either taking ART or receiving pre-ART care will be compared with each other and with that of HIV uninfected employees. There are no study visits associated with this study; all data will be collected from medical records maintained by the HIV/AIDS treatment program and the participants' employer. The financial costs and benefits of the treatment program for the participating company will also be estimated.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Employed by participating company for at least 1 year prior to study entry

Inclusion Criteria for Index Participants:

* Enrolled in the HIV/AIDS treatment program offered by the participating company

Exclusion Criteria for Index Participants:

* Enrolled in the HIV/AIDS treatment program prior to 01/01/04 or after 06/30/05

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: see elig
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-07-01 (Actual); Primary Completion 2005-07-01 (Actual); Study Completion 2005-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sydney B. Rosen, MPA, Principal Investigator — Boston University
Locations (1):
- Health Economics Research Office, Helen Joseph Hospital, Johannesburg, Gauteng, South Africa

REFERENCES:
- [Background] Fox MP, Rosen S, MacLeod WB, Wasunna M, Bii M, Foglia G, Simon JL. The impact of HIV/AIDS on labour productivity in Kenya. Trop Med Int Health. 2004 Mar;9(3):318-24. doi: 10.1111/j.1365-3156.2004.01207.x. PMID 14996359
- [Background] Rosen S, Vincent JR, MacLeod W, Fox M, Thea DM, Simon JL. The cost of HIV/AIDS to businesses in southern Africa. AIDS. 2004 Jan 23;18(2):317-24. doi: 10.1097/00002030-200401230-00023. PMID 15075551
- See also: Click here for the Program on the Social and Economic Impacts of the AIDS Epidemic Web site — http://sph.bu.edu/index.php?option=com_content&task=view&id=385&Itemid=485